CLINICAL TRIAL: NCT02570789
Title: A Proof of Concept Study to Evaluate the Use of Metabonomics and Lipidomics in Predicting Toxicity and Efficacy of Anti-VEGF Therapy in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Evaluation of Predictive Markers for Toxicity and Efficacy in Patients With mccRCC Treated by Anti-VEGF Therapy
Acronym: METASUN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough accrual
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UCL-ONCO 2012-09
Record Dates: First submitted 2015-09-17; First posted 2015-10-07 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with sunitinib or pazopanib (Experimental): This will be a non-randomized, proof-of-concept, prospective, longitudinal, multi-center study in patients with metastatic clear cell renal cell carcinoma with good or intermediate risk (based on MSKCC criteria) treated with sunitinib or pazopanib in first line.
  Interventions: Drug: patients with sunitinib or pazopanib

INTERVENTIONS:
Drug: patients with sunitinib or pazopanib — The treatment with sunitinib or pazopanib should comply with the recommendations written in the Belgian product information and the reimbursement criteria

SUMMARY:
The purpose of this study is to assess whether certain metabonomics and/or lipidomics features in correlation with pharmacokinetics before, during and after treatment with sunitinib or pazopanib in first line can predict toxicity and efficacy of sunitinib or pazopanib in metastatic clear cell renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man ≥ 18 Years old, histologically proven metastatic clear cell (or al least clear cell predominant) RCC,
* Good or intermediate risk according to MSKCC-criteria, Subjects falling into conditions for reimbursement of sunitinib or pazopanib in the context of mRCC,
* Measurable disease based on RECIST criteria (version 1.1) , Subject has given voluntary written informed consent,
* Subject is in the investigator's opinion, willing and able to comply with the protocol requirements, Subject has an ECOG ≤ 2,
* Subject with a life expectancy ≥ 3 months,
* Concurrent treatment with bisphosphonates and denosumab is allowed however it should have been started before screening of the study. If possible starting new medications between the baseline metabolo- and lipidomotype- and the first metabolo- and lipidomotypeanalysis should be avoided,
* Subjects having recovered from side effects from previous therapies to a grade 1 CTC vs 4.0 criteria

Exclusion Criteria:

* Patients with non-clear cell RCC and/or with sarcomatoid differentiation,
* Patients presenting any other type of cancer disease within 5 years from inclusion into this study; in the absence of cervical cancer or basocellular carcinoma, Patients with uncontrolled arterial hypertension,
* Patients with uncontrolled hypo- or hyperthyroidism,
* Patient had major surgery within 4 weeks before enrolment,
* Patient with myocardial infarction within 6 months prior enrolment or with NHYA class III otr IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia or electrocardiographic evidence of acute ischemia or active conduction system abnormalities,
* Patient has another serious medical condition that could potentially interfere with the completion of study,
* Sero-positive for HIV, Subject known to be hepatitis B surface antigen positive or who has an active hepatitis C infection,
* Subject has an active systemic infection requiring treatment,
* Female subject is pregnant or breast feeding, Subject enrolled in another clinical trial and/or receiving an investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2018-12 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment assessment by using RECIST 1.1 and adverse events will be documented using the NCI-CTC coding system (version 4.0) | up to 3 years

SECONDARY OUTCOMES:
Identifying the level metabolotype and/or lipidomotype of metastatic clear cell renal cell carcinoma patients before starting sunitinib or pazopanib (in comparison with healthy volunteers) on blood and urine samples by biochemistry techniques | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium